CLINICAL TRIAL: NCT05397808
Title: The Effects of Pilates Exercises on the Postpartum Period
Brief Title: Effects of Pilates Exercises on Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Bulguroglu, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Postpartum Disorder
Keywords: Pilates exercises; depression; sleep quality
MeSH Terms: conditions — Puerperal Disorders; Depression; Sleep Initiation and Maintenance Disorders | interventions — Exercise Movement Techniques; Respiration

STUDY DESIGN:
Intervention Model Description: Using a computer program, the investigators randomly placed individuals who completed the initial assessment into the pilates group or control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates group (Experimental): Pilates training will be held for eight weeks, two days a week for 1 hour. The investigators divided the individuals in the pilates exercise group into groups of 12 or 13 to verify whether they did the exercises correctly. A program including 15 minutes of warm-up, 30 minutes of Pilates exercises, and 15 minutes of cooling and stretching exercises was arranged for the pilates group. The activities were performed in ten repetitions. The exercise program recommended by the Australian Pilates and Physiotherapy Institute during postpartum will be used in the training.
  Interventions: Other: Pilates Training
- control group (Active Comparator): The control group was given breathing and relaxation exercises, which they would do two days a week for eight weeks, in the form of a home program. Diaphragmatic breathing and respiratory control were given as breathing exercises.
  Interventions: Other: breathing and relaxation exercises

INTERVENTIONS:
Other: Pilates Training — The group that received pilates training.
  Arms: pilates group
Other: breathing and relaxation exercises — The group who received breathing and relaxation exercises with a home program.
  Arms: control group

SUMMARY:
The postpartum period for the family is the period of adjustment in which a new order is established due to adding a new member to the family. For the mother, this period is a transitional period in which she has to adapt to her baby, postpartum disorders, the new order in the family, and changes in body image. Inactivity is common in today's world; increases the risk of various problems in new mothers. These problems negatively affect women's depression, functional level, sleep quality, and quality of life in the postpartum period. The Pilates method, developed by Joseph Pilates under the name of "Contrology," is the most well-known exercise method in the world for babies and mothers among today's exercise programs since it is an exercise method in which all systems, spirit, and body are integrated and coordinated, considering the whole physiological process.

This study aims to understand how depression, loss of functionality, sleep quality, functional levels, and quality of life levels of women who do pilates exercises with a physiotherapist are affected in the postpartum period.

DETAILED DESCRIPTION:
The investigators conducted the study at Ankara Medipol University, Faculty of Health Sciences, Department of Physical Therapy and Rehabilitation. This study was conducted by the principles set out in the Declaration of Helsinki. Fifty postpartum women aged 25-38 will be included in the study.

* Procedures The investigators assessed the participants by an experienced physiotherapist, who was blind to the randomization, at the start of the study and after the 8-week training. The group on which they depended was not disclosed to the participants until the end of the baseline evaluation. The investigators used a computer program for randomization and randomly placed individuals who completed the initial assessment into the pilates group (PG) or control group (CG). The investigators performed the Pilates exercises under the supervision of a certified physiotherapist with ten years of experience. The investigators asked the individuals not to inform the evaluator of their involvement in the training during the last evaluation. Before the study, the investigators explained the purpose and content of the survey to the participants and obtained written informed consent from all pregnant women to participate in the study.

Pilates training was done by an Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu lasted eight weeks, two days a week for one h. The investigators divided the individuals in the Pilates exercise group into two smaller groups of 12 or 13 to verify whether they correctly did the exercises. In this study, the investigators organized a program to include 15 min of warm-up, 30 min of Pilates exercises, and 15 min of cooling and stretching exercises. The exercises were done in 10 repetitions. The exercise program recommended by the Australian Pilates and Physiotherapy Institute during postpartum was used in training. During the Pilates exercises, investigators described the activities with different visual simulation techniques, and exercises were done together with Pilates breathing. The intensity of the exercises was increased by using different positions and elastic bands. The resistance was increased by starting with the red Therabant and switching to the blue band after two weeks. If the new resistance amount was challenging for the patient, the exercises were continued with the same color band for one more week. Stretching exercises and posture exercises were used during the cooling period. The subjects in the online pilates group were informed about side effects such as shortness of breath, dizziness, headache, muscle pain, and weakness. They were asked to stop exercising when there were any side effects.

-Statistical analysis The investigators will perform statistical analysis using SPSS software, version 21 (SPSS Inc. Chicago, IL, USA). The normal distribution of variables will be determined using histograms, probability plots, and a Shapiro-Wilk test. Because of an abnormal distribution, median and interquartile range (IQR) were used for descriptive statistics. Numerical variables showing normal distribution were shown as mean±standard deviation. The investigators will use a Mann-Whitney U test to compare baseline and change values between groups. The investigators will use Wilcoxon Test to compare baseline values within the group and values after eight weeks. The significance level will be set at p < 0.05 for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal birth
* First birth
* At least six weeks postpartum
* Absence of any anomaly in the mother or baby after birth
* Being between the ages of 25-38
* Having a body mass index <30

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems that may affect the results of the research.
* Participating in other exercises or physiotherapy programs during the past 6 months.
* Cesarean delivery

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Depression- Baseline | Baseline
  Edinburgh Postpartum Depression Scale (EPDS) is a self-report scale consisting of 10 items, in a 4-point Likert format. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point for EPDS is 13 points. Accordingly, 13 points and above indicate the risk of depression.
Depression- Post intervention | Assessment will be conducted immediately after the intervention
  Edinburgh Postpartum Depression Scale (EPDS) is a self-report scale consisting of 10 items, in a 4-point Likert format. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point for EPDS is 13 points. Accordingly, 13 points and above indicate the risk of depression.
Oswestry Disability Index- Baseline | Baseline
  The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, degree of pain change, travel, and social life. When calculating the total score, it is multiplied by two and expressed as a percentage. The maximum score is "100," and the minimum score is "0". As the total score increases, the level of disability also increases.
Oswestry Disability Index- Post intervention | Assessment will be conducted immediately after the intervention
  The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, degree of pain change, travel, and social life. When calculating the total score, it is multiplied by two and expressed as a percentage. The maximum score is "100," and the minimum score is "0". As the total score increases, the level of disability also increases.
Postpartum Sleep Quality Scale- Baseline | Baseline
  The PSQS is scored using a 5-point Likert scale ranging from 0 to 4 (0 = never,1= rarely,2= sometimes,3= often, and 4 = always). The items with an asterisk are scored in reverse order. Possible scores for the PSQS range from 0 to 56, with no cutoff point designated and higher scores indicating poor sleep quality.
Postpartum Sleep Quality Scale- Post intervention | Assessment will be conducted immediately after the intervention
  The PSQS is scored using a 5-point Likert scale ranging from 0 to 4 (0 = never,1= rarely,2= sometimes,3= often, and 4 = always). The items with an asterisk are scored in reverse order. Possible scores for the PSQS range from 0 to 56, with no cutoff point designated and higher scores indicating poor sleep quality.
The Inventory of Functional Status After Childbirth- Baseline | Baseline
  The IFSAC consists of five subscales, including five dimensions of functional status and 36 four-point Likert-type questions to determine postpartum recovery. Each question of the IFSAC has been evaluated over four points (from one to four). A high score (close to four) indicates high functional status.
The Inventory of Functional Status After Childbirth- Post intervention | Assessment will be conducted immediately after the intervention
  The IFSAC consists of five subscales, including five dimensions of functional status and 36 four-point Likert-type questions to determine postpartum recovery. Each question of the IFSAC has been evaluated over four points (from one to four). A high score (close to four) indicates high functional status.
Maternal Postpartum Quality of Life Questionnaire- Baseline | Baseline
  Postpartum quality of life is a scale that is evaluated according to the perception of the mother and consists of five sub-dimensions and a total of 40 items. The scores obtained after the procedure are summed up and divided by the number of scale questions (40 items), and a fixed value (15) is added to the number obtained from the section to avoid negative results, and the result is found. Thus, the Quality of Life Scores is in the range of 0-30. The higher the score obtained from the scale, the higher the person's postpartum quality of life, and lower scores indicate a lower postpartum quality of life.
Maternal Postpartum Quality of Life Questionnaire- Post intervention | Assessment will be conducted immediately after the intervention
  Postpartum quality of life is a scale that is evaluated according to the perception of the mother and consists of five sub-dimensions and a total of 40 items. The scores obtained after the procedure are summed up and divided by the number of scale questions (40 items), and a fixed value (15) is added to the number obtained from the section to avoid negative results, and the result is found. Thus, the Quality of Life Scores is in the range of 0-30. The higher the score obtained from the scale, the higher the person's postpartum quality of life, and lower scores indicate a lower postpartum quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: HALİL I BULGUROGLU, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Altındağ, Ankara, Turkey (Türkiye)